CLINICAL TRIAL: NCT04548570
Title: Closure vs Non Closure of Rectus Muscle at Cesarean Section Reducing Post Cesarean Adhesions
Brief Title: Closure vs Non Closure of Rectus Muscle at Cesarean Section 5 Year Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany saad, assisstant professor, Cairo University
Other Study IDs: assisstant professor
Record Dates: First submitted 2020-05-19; First posted 2020-09-14 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Intraperitoneal Adhesions After Rectus Muscles Approximation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- approximation of both recti group
  Interventions: Procedure: approximation of both rectus muscles
- non approximation of both recti group
  Interventions: Procedure: approximation of both rectus muscles

INTERVENTIONS:
Procedure: approximation of both rectus muscles — closure of both rectus muscle before closure of rectus sheeth

SUMMARY:
approximation of both recti during lower segment cesarean section may be an important step to lower incidence of intraabdominal adhesions . peritoneal adhesions are of major medical importance and are associated with clinical problems such as chronic pain and infertility.

DETAILED DESCRIPTION:
all patients included in the study should be had the operative history of the previous cesarean section and were done in the cairo university and divid them into 2 groups. 1st group were both recti approximated while the second group were closed without approximating both recti. all patients will be subjected to lower segment cesarean segment to assess the intraperitoneal adhesions, mean operative time, mean hospital stay, postoperative distension, bowel sounds, postoperative infections and morbidity

ELIGIBILITY:
Inclusion Criteria:

* all patients of first lower segment cs at kasr al ainy with previous recorded data including operative data, postoperative data including complications. all patients included in the study are elective cesarean section at 38 weeks of gestation

Exclusion Criteria:

* no history of infection or medical disease
* no history of previous laparotomies
* no history of pregnancy complications
* patients noted to have intraperitoneal adhesions in first cesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients who will subjected to cesarean section with history of previous cesarean section in the same hospital with operative notes and techniques
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
assessment of the intraperitoneal adhesions post rectus muscle closure | intraoperative
  assessment of adhesions bands between the pelvic organs and bowel

SECONDARY OUTCOMES:
mean operative time | intraopertive time
  calculate the mean time for closure of both recti
mean hospital stay | posoperative within first 48 hrs
  assess the postoperative time of hospital stay
mean postoperative bowel sounds | posoperative within 24 hrs
  interval between operation and listening the bowel sounds
postoperative distension | posoperative within 24 hrs
  assessment of bowel distension postoperative
postoperative morbidity and infections | posoperative within 1 week
  assess the tempreture, scars

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt